CLINICAL TRIAL: NCT06856551
Title: Using Tailored Messages to Encourage Healthy Lifestyle Choices in a Brief, Self-directed Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Florida (Other)
Responsible Party: Principal Investigator, Paul Fuglestad, Associate Professor, University of North Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 724308
Record Dates: First submitted 2025-02-14; First posted 2025-03-04 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-02

CONDITIONS: Weight Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Minimal contact control (Active Comparator): Participants in the control group received a pamphlet about general dietary and physical activity guidelines.
  Interventions: Behavioral: Minimal contact control
- Promotion focus group (Experimental): Participants completed a 1-hour educational information session with study staff and received a packet which contained information about energy balance, healthy food choices, exercise recommendations, strategies for weight control, goal setting, and responding to lapses. Participants were encouraged to track their food intake and exercise with a provided log book or free apps (Lose It!; MyFitnessPal). All messages and study tasks were framed in terms of promotion focus. Email messages were sent every 2 to 3 weeks to reinforce the study messages about health promotion and weight control.
  Interventions: Behavioral: Promotion and Prevention Interventions
- Prevention focus group (Experimental): Participants completed a 1-hour educational information session with study staff and received a packet which contained information about energy balance, healthy food choices, exercise recommendations, strategies for weight control, goal setting, and responding to lapses. Participants were encouraged to track their food intake and exercise with a provided log book or free apps (Lose It!; MyFitnessPal). All messages and study tasks were framed in terms of prevention focus. Email messages were sent every 2 to 3 weeks to reinforce the study messages about health promotion and weight control.
  Interventions: Behavioral: Promotion and Prevention Interventions

INTERVENTIONS:
Behavioral: Minimal contact control — Participants in the control group received a pamphlet about general dietary and physical activity guidelines.
  Arms: Minimal contact control
Behavioral: Promotion and Prevention Interventions — regulatory focus groups, participants completed a 1-hour educational information session with study staff and received a packet which contained information about energy balance, healthy food choices, exercise recommendations, strategies for weight control, goal setting, and responding to lapses. Participants were encouraged to track their food intake and exercise with a provided log book or free apps (Lose It!; MyFitnessPal). The informational content and intervention procedures were identical except for the framing of messages and tasks. The prevention messages emphasized protecting one's health (e.g., failing to regularly exercise can undermine your weight control program and lead to poor health; if you do not vigilantly follow these behaviors, you will not fulfill your weight control goals or protect your health and well-being; not eating fruits and vegetables results in failure to supply the body with the nutrients it needs). The promotion messages emphasized promoting one's health
  Arms: Prevention focus group; Promotion focus group

SUMMARY:
The study aimed to investigate 1) if a brief, regulatory focus-based intervention could promote weight control and changes in certain lifestyle behaviors and 2) how weight was affected by changes in these behaviors. The lifestyle behaviors of interest included meal regularity, self-monitoring of diet and physical activity, fast-food eating, screen related viewing and eating, dietary modifications, self-weighing, and physical activity. It was hypothesized that increases in meal regularity, self-monitoring, healthy dietary modifications, self-weighing, and physical activity would lead to better weight control over six months. Conversely, it was hypothesized that increases in fast food consumption and screen related eating and viewing would lead to poorer weight control over six months. It was expected that promotion and prevention conditions, relative to the control condition, would lead to better weight control and increases in meal regularity, self-monitoring, healthy dietary modifications, self-weighing, and physical activity, and decreases in fast food consumption and screen related eating and viewing. Furthermore, it was expected that the promotion condition would lead to better outcomes than the prevention condition.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* generally healthy
* BMI between 18.5 and 35

Exclusion Criteria:

* pregnancy within the past 6 months
* current pregnancy
* plan to get pregnant in the next 6 months
* serious physical or psychological problems that would contraindicate participation in a weight-related program
* history of anorexia or bulimia
* diabetes or hypertension
* current participation in a weight-loss program
* BMI < 18.5, >35.0

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-10-30 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
Weight Change | baseline, 3 months, 6 months
  Participant were weighed by study staff during a baseline measurement session (M = 153.7 lb, SD = 31.6) and then again after 6 months (M = 149.9 lb, SD = 28.9). Weight was self-reported at 3 months (M = 150.7 lb, SD = 29.4).

SECONDARY OUTCOMES:
meal regularity change | baseline, 3 months
  Participants were asked about the number of times in a typical week they 1) ate breakfast, 2) ate lunch, and 3) ate dinner. They responded on a 5-point scale: 0 times, 1-2 times, 3-4 times, 5-6 times, or 7+ times. Mean scores were created for the baseline measurement session (M = 4.00, SD = .73) and for the 3-month measurement session (M = 4.17, SD = .72).
fast-food eating change | baseline, 3 months
  Participants were asked about the number of times in a typical week they 1) ate food prepared at a fast-food restaurant and 2) purchased food at a convenience store/ gas station. They responded on a 5-point scale: 0 times, 1-2 times, 3-4 times, 5-6 times, or 7+ times. Mean scores were created for the baseline measurement session (M = 1.74, SD = .66) and for the 3-month measurement session (M = 1.63, SD = .53).
screen related eating and viewing change | baseline, 3 months
  Participants indicated the frequency per week that they 1) ate a meal while watching TV, 2) ate a snack while watching TV, and 3) ate after 8 pm. The participants responded by using a 5-point scale: 0 times, 1-2 time, 3-4 times, 5-6 times, or 7+ times. They also indicated the number of hours on an average day that they 4) use a phone/tablet/computer, 5) watch TV and 6) sit or recline (not including sleeping). Their responses were recorded on a 7-point scale: 0, <1 hour, 1 hour, 2 hours, 3 hours, 4 hours, or 5+ hours. Mean scores across the six items were calculated for the baseline measurement session (M = 3.44, SD = .90) and the 3-month measurement session (M = 3.34, SD = .90).
dietary modifications change | baseline, 3 months
  Dietary modification was measured by asking participants how often they 1) reduced/limited their portions, 2) decreased/limited snacks, 3) decreased/limited sweets, 4) decreased/limited fried food, 5) decreased/limited carbs, 6) decreased/limited fat, 7) ate fruits and vegetables, and 8) planned meals. Participants responded on a 5-point scale: never, rarely, sometimes, often, or very often. Mean scores were calculated for the baseline measurement session (M = 2.96, SD = 0.74) and for the 3-month measurement session (M = 3.32, SD = 0.73).
self-monitoring change | baseline, 3 months
  For self-monitoring, participants were asked how often they wrote down the calorie content of the foods they ate and the amount and types of exercise they did. Participants responded on a 5-point scale: never, rarely, sometimes, often, or very often. Mean scores were then calculated for the baseline measurement session (M = 1.86, SD = 1.03) and for the 3-month measurement session (M = 2.85, SD = 1.26).
self-weighing change | baseline, 3 months
  At baseline, participants responded to the question "How often do you weigh yourself?" on a 7-point scale: never, about once a year or less, every couple of months, every month, every week, every day, or more than once a day (M = 3.83, SD = 1.31). At 3 months, they responded to the question "In the past week, how many times did you weigh yourself?" on a 5-point scale: never, 1-2 times, 3-4 times, 5-6 times, or 7 or more times (M = 2.01, SD = 1.02).
physical activity change | baseline, 3 months
  To measure physical activity, participants were asked how often they 1) planned their exercise, 2) walked for at least 30 minutes at a time, and 3) engaged in other moderate to vigorous exercise. Participants responded on a 5-point scale: never, rarely, sometimes, often, or very often. Mean scores were calculated for the baseline measurement session (M = 3.31, SD = .94) and for the 3-month measurement session (M = 3.55, SD = 1.08).

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Will be shared on open science framework.